CLINICAL TRIAL: NCT07126340
Title: The Effect of Foot Massage on Pain, Satisfaction, and Analgesic Consumption in Patients Undergoing Total Knee Arthroplasty
Brief Title: Effect of Foot Massage on Pain and Analgesic Consumption in Total Knee Prosthesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alev Keskin (Other)
Responsible Party: Sponsor-Investigator, Alev Keskin, RN, MSc Nurse, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Alev Keskin
Record Dates: First submitted 2025-04-26; First posted 2025-08-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Cold Therapy; Total Knee Arthroplasty; Postoperative Pain; Foot Massage; Analgesic Consumption
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of Foot Massage and Cold Application on Postoperative Pain (Active Comparator): The cold application protocol will be initiated upon the patient's arrival at the clinic after surgery. Cold therapy will be applied for 20 minutes every two hours and will continue for 48 hours postoperatively. In addition to cold therapy, patients will receive foot massage performed according to a standard technique. The massage will include effleurage (stroking and gliding), petrissage (kneading), and friction maneuvers. Vaseline will be used during the massage to minimize skin friction and facilitate smooth hand movements.
  Interventions: Other: Foot Massage and Cold Application
- Effect of Cold Application on Postoperative Pain (Active Comparator): The cold application protocol will be started from the moment the patient comes to the clinic after surgery. Cold application will be done for 20 minutes and every 2 hours. This application will be continued for the patient for 48 hours from the postoperative period.
  Interventions: Other: Cold Application

INTERVENTIONS:
Other: Foot Massage and Cold Application — The patient will receive both cold application and foot massage after total knee arthroplasty.
  Arms: Effect of Foot Massage and Cold Application on Postoperative Pain
Other: Cold Application — After total knee arthroplasty, the patient will receive routine cold application.
  Arms: Effect of Cold Application on Postoperative Pain

SUMMARY:
This randomized controlled trial aims to examine the effects of foot massage combined with cold application on postoperative pain, patient satisfaction, and analgesic consumption in individuals undergoing Total Knee Arthroplasty (TKA). The study will be conducted in the Orthopedics and Traumatology Department of Çukurova University Balcalı Hospital, which includes an 18-bed orthopedic unit.

Eligible patients will be randomly assigned to either the intervention group or the control group.

* Intervention group: Patients will receive both cold application and foot massage. Cold therapy will be administered for 20 minutes every 2 hours for the first 48 hours postoperatively. Foot massage will be performed twice daily (morning and evening) for two days following drain removal, using standardized massage techniques.
* Control group: Patients will receive only cold application following the same schedule and procedure as the intervention group.

Data will be collected using the Patient Information Form, the Short Form of the Brief Pain Inventory, the Numeric Rating Scale, and the Newcastle Satisfaction with Nursing Care Scale. Statistical analyses will be conducted using SPSS, and findings will be interpreted at a 95% confidence level (p < 0.05).

Ethical approval has been granted by the Çukurova University Non-Interventional Clinical Research Ethics Committee. Institutional permission will be obtained prior to data collection. Participation will be voluntary, and all data will be treated confidentially.

ELIGIBILITY:
Inclusion Criteria

* Being 18 years or older
* Ability to speak Turkish
* No visual or hearing impairment
* No cognitive disability
* Undergoing unilateral knee replacement surgery
* Volunteering to participate in the study

Exclusion Criteria

* Presence of any intellectual disability or psychiatric disorder
* History of diabetes
* Presence of neurological or cerebrovascular disease
* Diagnosis of deep vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale, | One minute
  The patient is asked to choose the number that best reflects the pain intensity, 0=no pain, 10= equal to the worst (unbearable) pain.
Brief Pain | Five minutes
  The inhibition of individuals' daily living activities due to pain experienced in the last 24 hours is similarly assessed using a numerical scale (0 = not affected at all, 10 = completely affected).

SECONDARY OUTCOMES:
Newcastle Nursing Satisfaction Scale | Ten minutes
  The evaluation of all the items marked on the scale is converted to 100 after the pu moments are collected and made over 0-100 points. The fact that the total score is 100 indicates that all dimensions of nursing care are satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova Üniversitesi, Adana, University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No